CLINICAL TRIAL: NCT05027789
Title: Compensation Training and Lifestyle Modifications to Promote Healthy Aging in Persons at Risk for Alzheimer's Disease: a Digital Application Supported Intervention (Brain Boosters 2)
Brief Title: Brain Boosters 2 in Persons at Risk for Alzheimer's Disease: a Digital Application Supported Intervention
Acronym: BB2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1764579; 1R01AG066748-01A1 (NIH)
Record Dates: First submitted 2021-08-05; First posted 2021-08-30 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Memory Disorders; Cognitive Impairment
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This project will utilize a randomized controlled trial (RCT) design with single blinding (outcomes examiner) comparing the structured intervention (combined structured training in compensation and lifestyle modification, assisted by the EMMA) to the self-guided intervention group, which focuses on providing education and allowing participants to choose how to implement the information was chosen to account for the impact of two general factors: 1) the provision of information, and 2) the social support and stimulation provided by attending a group-based intervention.
Who Masked: Outcomes Assessor
Masking Description: The outcomes examiner will be blinded to participants' study arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Guided Group (Active Comparator): Subjects in this group will be provided education on memory support strategies and healthy lifestyles. Participants will decide how they want to implement this information into their daily lives. The study will also provide information on various commercially available digital and other tools that might help participants implement healthy changes their lives. One in every three participants will be enrolled in this group (selected randomly).
  Interventions: Behavioral: Self-Guided
- Structured Group (Active Comparator): Subjects in this group will will be provided with specific recommended behavior targets (e.g., like how much exercise you should engage in each week). Participants will also receive an iPad to use throughout the study and follow up period with the digital application installed. Subjects will be asked to use the digital application to record their activity and to receive reminders to complete this information. Two in every three participants will receive the iPad and digital application. Participants in this group will receive training on how to use the digital application. The researchers can install the digital application on the subjects' personal iPad or smartphone if they prefer.
  Interventions: Behavioral: Structured Group

INTERVENTIONS:
Behavioral: Self-Guided — People in this arm will come to 15 information sessions. These sessions will provide training and education on memory support strategies and healthy lifestyles. You will decide how you want to implement this information into your daily life.
  Arms: Self-Guided Group
Behavioral: Structured Group — People in this group will come to 15 information sessions. The study will provide recommended behavior targets (like how much exercise you should have each week). Participants in this group will either receive an iPad or have a special application installed on their own personal device. They will receive training on how to use the application, and will be asked to use the application to record their activities and receive reminders.
  Arms: Structured Group

SUMMARY:
The purpose of this research is to determine if training in memory support aids and healthy lifestyle activities (physical exercise, mentally stimulating activities and stress management) can have a positive effect on memory, thinking, and activities that people do every day. Participation in this study will involve being placed into one of two groups: a Self-Guided Intervention Group or a Structured Intervention Group. Both groups will be asked to attend group sessions in which they will be provided education on memory support strategies and lifestyle changes. The Structured Intervention Group will also be provided with an iPad and a digital application (called EMMA) to track their activity. Study participation involves a 6-month intervention and completing outcome measures at 4 different time points for up to a year.

DETAILED DESCRIPTION:
Participants in this research will be asked to participate in group sessions about memory support strategies and healthy behaviors. They may also choose to have a partner participate in this study with them, but it is not required.

There will be weekly sessions for 10 weeks, followed by sessions 1 to 2 times per month for the next 4 months.

Participants will be asked to complete healthy lifestyle activities on their own. Before the intervention starts and at three time points after the intervention, we will collect cognitive assessments and questionnaires to measure the possible impact of the treatment. The post-intervention assessments will take place right after completion of the intervention, and then 6 and 12 months later.

Before the start of the study, participants will be required to get permission from their primary care provider to ensure that it is safe for them to complete physical aerobic exercise.

The Self-Guided and Structured Intervention Groups will be required to participate in the following study activities:

Intervention Training Sessions:

Participants will be asked to attend 15 information sessions that include:

1. training on ways to help support memory like remembering appointments or taking medication and
2. training on increasing interest in three health behaviors known to reduce risk of memory declines (physical exercise, mental stimulation, stress management).

These sessions will be in a group of up to 15 people and will last about 2 hours each. For 10 weeks, there will be sessions every week, and then for the next 4 months there will be 1-2 session each month.

There are two different versions of the intervention we are evaluating. Participants will be randomly assigned into one of the two groups. Both groups provide similar information about memory support strategies and lifestyle modifications to promote cognitive health.

Self-Guided Group

Participants in the self-guided group will:

* Receive education on memory support strategies and healthy lifestyles.
* Decide how they want to implement this information into their daily life.
* Receive information on various commercially available digital and other tools that might help them implement healthy changes in their life.
* The chance that participants will be in this group is random, like flipping a coin. One in every three participants will be enrolled in this group.

Structured Group

Participants in this group will:

* Receive specific recommended behavior targets (e.g., like how much exercise they should engage in each week).
* Receive an iPad to use throughout the study and follow up period with the digital application installed.
* Be asked to use the digital application to record their activity and to get reminders to complete this information.

Two in every three participants will receive the iPad and digital application.

Participants in this group will receive training on how to use the digital application.

Participants with their own iPad and/or smartphone can install the digital application on their personal iPad or smartphone if they prefer.

Both the Self-Guided and Structured groups will complete the following assessments:

Physical Assessment:

Cardiovascular health - This questionnaire will ask about age, sex, education, blood pressure, total cholesterol level, body-mass index and complete a short test of physical activity.

Cholesterol Test:

A blood test at the University of California Davis Pathology laboratory will be performed for any participant who has not had this test in the past year. Participants must fast overnight and have nothing but water for 12 hours before the blood test. Approximately 4 milliliters (or about 1 teaspoon) of blood will be drawn for this test.

Memory and Behavior Questionnaires:

Tests of memory and thinking and questionnaires about health and behaviors will be completed at the beginning of the study and three additional times (every 6 months). Study partners will also be asked to complete some questionnaires about the participant.

Participants who are randomized to the Structured Intervention Group will also be asked to complete these additional assessments:

* Week-Long Assessment:

  o Structured Intervention Group participants will be asked to complete daily assessments for one week at four different times during participation. This will include questions about the experience with EMMA and some short memory and thinking assessments.
* Digital application (EMMA) Experiences Interview:

  * A subset of participants in the Structured Intervention Group will be asked to complete an interview about their experience with using EMMA. This interview will occur over the telephone or video conferencing (such as Zoom) and will be recorded for scoring and quality assurances. The researchers will keep these recordings until the study is complete (about 5 years). This is completely voluntary, and participants can choose not to complete the interview.

ELIGIBILITY:
Inclusion Criteria:

* The target population is cognitively normal older adults with Subjective Cognitive Concerns (SCC). SCC will be operationalized as

  1. a positive complaint in response to the question: 'Have you experienced a decline in your memory or other aspect of thinking in the last 1-3 years that seems worse than others of your age'
  2. normal cognition on the modified Telephone Interview of Cognitive Status (mTICS)
  3. independent function in daily life.
* Age 65 or older
* English speaking
* Lower level of engagement in healthy lifestyle behaviors and compensation use at study baseline (i.e., broadly defined as not a regular exerciser)
* Approval from primary care (due to physical exercise component of the intervention)
* Open to utilizing digital tools such as a digital calendar in daily life

Exclusion Criteria:

* Known diagnosis of dementia or cognitive impairment;
* Other known neurological condition with potential to affect cognition (e.g., Parkinson's disease)
* Reported history of severe psychiatric disorder (e.g., self-reported history of bipolar disorder or schizophrenia or other psychotic disorder)
* Inability to complete the study protocols due to severe vision or hearing difficulties.
* Has previously participated in a previous version of Brain Boosters, or another study utilizing the Digital Memory Notebook (DMN) application or EMMA.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 263 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Logical Memory | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  A standardized assessment of narrative episodic memory.
Free and Cued Selective Reminding Test (FCRT) | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  A standardized assessment of immediate and delayed memory by using cues or free recall
Digit Span | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  A standardized assessment of attention and working memory by recalling short lists of numbers immediately in either forward or backwards order.
Trail Making | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  A standardized assessment of executive functioning by assessing following order but switching between letters and numbers.
Digit Symbol | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  A standardized assessment of executive functioning by having participants match symbols and letters.
Verbal Fluency | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  A standardized assessment of executive functioning by having participants list as many words they can that start with a specific letter.
Royal Prince Alfred Prospective Memory Test | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  A standardized assessment of prospective memory by asking participants to remind the examiner of a task at different intervals throughout the session.
Everyday Function | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  Evaluates participants everyday cognition through a variety of self-report questions about their daily functioning.

SECONDARY OUTCOMES:
Coping Self efficacy (CSES) | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  Questionnaire measuring perceived self-efficacy for coping with challenges and threats
Center for Epidemiologic Studies Depression Scale (CES-D) | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  Self-report measure of depression
Perceived Stress Scale (PSS) | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  Self-report measure of stress
Satisfaction with Life | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  Self-report measure of life satisfaction
Purpose in Life | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  Self-report measure of life purpose
Short Physical Performance Battery | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  Measures gait speed, balance and sit to stand
Brief Resiliency Scale (BRS) | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  Self-reported measure of resilience
Patient Reported Outcomes Measurement Information System (PROMIS) General Health and Quality of Life Measure | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  two question scale assessing feelings on general health and quality of life.
Cooperative Study Activities of Daily Living (ADL) Prevention Instrument (ADCS-ADL-PI) | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  questionnaire measuring functional abilities (e.g., managing finances, medication, shopping, laundry)
Everyday Compensation (EComp) | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  Questionnaire measuring the behavioral compensatory strategies in the context of performing tasks like managing finances, medication, shopping, laundry, etc.
Community Healthy Activities Model Program for Seniors (CHAMPS) | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  Questionnaire measuring frequency and duration of various physical activities and cognitively stimulating activity
Positive Affect and Negative Affect Scale (PANAS) | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  Questionnaire measuring of positive and negative affect
The Gratitude Questionnaire - Six Item Form | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  Questionnaire measuring the frequency of feelings of gratitude
Mindfulness Inventory | Change in assessment scores from baseline to 6-months, 12-months, and 18-months
  Questionnaire measuring the construct of mindfulness in daily life (e.g. being aware of thoughts and feelings as well as external events).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Farias, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Alzheimer's Disease Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tomaszewski Farias S, Fox J, Dulaney H, Chan M, Namboodiri S, Harvey DJ, Weakley A, Rahman S, Luna C, Beech BF, Campbell L, Schmitter-Edgecombe M. Memory support training and lifestyle modifications to promote healthy aging in persons at risk for Alzheimer's disease: a digital application supported intervention (Brain Boosters). BMC Geriatr. 2023 Dec 21;23(1):881. doi: 10.1186/s12877-023-04574-x. PMID 38129775